CLINICAL TRIAL: NCT05346770
Title: Pharmacist-led Interventions to Improve Medication Use: Series of Case-reports
Brief Title: Pharmacist-led Interventions to Improve Medication Use
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: TRHC-CS-2021-001
Record Dates: First submitted 2022-03-02; First posted 2022-04-26 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Pharmacogenomics; Old Age
MeSH Terms: interventions — Behavior Therapy; Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individual Patient: Each case will represent one individual patient and patient case. The cases may not be related and may cover different clinical practice areas.
  Interventions: Behavioral: Behavioral Intervention; Diagnostic Test: Diagnostic Test; Other: Data Analysis

INTERVENTIONS:
Behavioral: Behavioral Intervention — A behavioral intervention could include changing the time of day a drug is taken.
Diagnostic Test: Diagnostic Test — A patient may receive a pharmacogenomic test via cheek swab to find PGx results. This is a benign intervention with little to no risk to the patient.
Other: Data Analysis — Medication safety reviews, and retrospective or prospective data analysis may occur as a result of participation in a case study.

SUMMARY:
The objective of this project is to stimulate identification and report of patient's medical story for whom their clinical conditions beneficiated from pharmacists' interventions based on a medication safety review. Cases will be systematically identified and reported in the scientific (peer review journals) and clinical communities in order to inform and provide better care.

DETAILED DESCRIPTION:
METHODS TRHC aims to collect data about participants using direct or retrospective observations such as patient's demographics, medical lab tests, clinical decision support systems, and examination of medical records and drugs. Specific case studies could include medication safety reviews, behavioral interventions, pharmacogenomic testings (PGx), and prospective or retrospective analyses of a patient's drug regimen, or medical records. Case reports covered under this protocol will be limited to single case reports.

TRHC pharmacists will maintain their routine health care practices. TRHC clinical research scientists and/or pharmacy residents will provide assistance and guidance. The writing process will be performed and supervised by TRHC scientist researchers.

Setting and Practice Description TRHC, d/b/a CareKinesis, is the first national pharmacy that provides science-based medication risk identification and mitigation technologies and services. CareKinesis utilizes medication decision support tools and pharmacists certified in geriatrics to provide pharmacy services for various healthcare organizations including PACE organizations (described above). Presently, CareKinesis services more than 35 PACE organizations, including approximately 100 PACE sites, across the United States. As a national PACE pharmacy provider since 2011, CareKinesis focuses on improving medication regimens to reduce medication-related risks while enhancing economic, clinical and humanistic outcomes. Pharmacist-led PGx clinical services and medication safety reviews are currently being offered to PACE organizations under the direction of licensed healthcare prescribers by TRHC (CareKinesis). In addition, TRHC provides risk stratification and medication safety review for non-PACE organizations and national health plans to identify trends in medication prescribing, and healthcare expenditures by risk level. This allows TRHC (CareKinesis) to assess large populations throughout the United States to validate the MedWise® clinical decision support system.

Each case report will be limited to a single patient.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all the following criteria will be considered:

1. Patient enrolled in a healthcare organization where TRHC provides pharmacy services during the implementation period.
2. Patient (or legal representative) able to understand, and provide informed consent to publish his/her case story.
3. Patient's case will provide generalizable knowledge to the existing literature based on direct observation, interview, benign behavioral intervention, or findings from drug regimen or drugs claims data.

Exclusion Criteria:

Patients with one of the following criteria will be excluded:

a) Patient's refusal to participate in a case study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient enrolled in a healthcare organization where Tabula Rasa Healthcare provides pharmacy services during the implementation period.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-01-24 (Estimated); Study Completion 2024-07-24 (Estimated)

PRIMARY OUTCOMES:
Medication safety reviews of patient drug regimen characteristics will be conducted to determine potential drug-drug interactions. | 1 year
  Medication safety reviews will be conducted and reported using Tabula Rasa Healthcare proprietary software MedWise to assign a Medication Risk Score. This evaluation incorporates over-the-counter medications, herbals, and supplements to illuminate simultaneous, multi-drug interactions. Based on the data, patients are assigned a risk score ranging from 0 to 50, where 0-9 indicates minimal risk, 10-14 indicates low risk, 15-19 indicates intermediate risk, 20-29 indicates high risk, and 30 and above indicates severe risk.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, PhD, Principal Investigator — TRHC
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.cdc.gov/nchs/products/databriefs/db328.htm#Summary.